CLINICAL TRIAL: NCT02069561
Title: Effects of Eicosapentaenoic Acid on Molecular, Metabonomics and Intestinal Microbiota Changes, in Subjects With Long-standing Inflammatory Bowel Disease
Brief Title: Effects of Eicosapentaenoic Acid on Subjects at High Risk for Colorectal Cancer
Acronym: EPAUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Luigi Ricciardiello, Associate Professor of Gastroenterology, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EPAUC/2013
Record Dates: First submitted 2014-02-19; First posted 2014-02-24 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Eicosapentaenoic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eicosapentaenoic Acid (Experimental): Subjects with long-standing ulcerative colitis and meeting the inclusion criteria will receive 2 g/day of Eicosapentaenoic Acid as a supplement for 90 days
  Interventions: Dietary Supplement: Eicosapentaenoic Acid
- Normal controls (No Intervention): Five patients undergoing screening colonoscopy and polypectomy using biopsy forceps. Six biopsies of healthy mucosa will be collected at the time of colonoscopy. Faeces, urine and blood samples will be collected prior to performing colonoscopy. The samples will serve as healthy reference for the basic studies.

INTERVENTIONS:
Dietary Supplement: Eicosapentaenoic Acid — Twenty patients with long-standing ulcerative colitis undergoing the usual colonoscopic surveillance + biopsy sampling will be recruited. At entry six extra biopsy samples will be collected from the colon. We will also collect blood (for serum, plasma and red cells isolation), urine and stools. Subjects will then receive 2 g/day of Eicosapentaenoic Acid (ALFA ™, SLA Pharma AG, Switzerland) as a supplement for 90 days. At the end of the study each subject will undergo sigmoidoscopy for the collection of 6 biopsies. Blood, urine and stools will be obtained prior to the procedure.
  Other Names: ALFA ™
  Arms: Eicosapentaenoic Acid

SUMMARY:
The aim of this study is to test Eicosapentaenoic acid's effects on markers relevant to colorectal carcinogenesis, RNA and DNA profiles, and the possibility that Eicosapentaenoic Acid treatment might be associated with changes of the gut microbiota and metabolomic profiles in patients with long-standing ulcerative colitis.

ELIGIBILITY:
Arm: experimental

Inclusion Criteria:

* Patients with ulcerative colitis (diagnosed based on clinical criteria, endoscopic and histological) lasting over 8 years, with no clinical activity (SCCAI = 0), and in stable treatment (without any change in treatment in the previous 3 months) with mesalamine, immunomodulators and / or biologics.
* Baseline fecal calprotectin> 150 micrograms / g.
* Signed informed consent.

Exclusion Criteria:

* Patients receiving systemic steroids in the two months prior to study entry.
* Patients taking concomitant warfarin or other blood thinners.
* Known or suspected hypersensitivity to eicosapentaenoic acid/omega 3.
* Women who are pregnant or of childbearing age who do not accept the use of contraceptive methods specified in the study (oral contraception, IUDs) and breastfeeding women.
* Patients with severe medical conditions that, in the opinion of the investigator, contraindicate the patient's participation in the study.
* Changes of treatments and / or use of experimental drugs within 3 months before inclusion in the study.
* Use of Probiotics

Arm: no intervention

Inclusion criteria

* Subjects undergoing screening colonoscopy within the regional colorectal cancer screening programme
* Signed informed consent
* Polypectomy with biopsy forceps.

Exclusion criteria

* HBV-positive, HCV-positive, HIV-positive or otherwise affected by infectious diseases
* Subjects undergoing chemo and radiation therapy within six months prior to surgery
* Patients receiving systemic steroid in the two months prior to study entry
* Patients undergoing antibiotic therapy within three months prior to the study
* Patients treated with probiotics

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Changes of RNA profiles (gene expression and micro RNA) from baseline | baseline and at 3 months
Changes of DNA methylation profiles | baseline and 3 months
Changes in cell proliferation | baseline and 3 months
Changes of apoptosis | baseline and 3 months

SECONDARY OUTCOMES:
Changes of circulating cytokines from baseline | baseline and 3 months
Changes of membrane fatty acid composition from baseline | baseline and 3 months
Changes of metabolomic profiles from baseline | baseline and 3 months
Change of Microbiota composition from baseline | baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Ricciardiello, MD, Principal Investigator — Azienda Ospedaliero Universitaria Policlinico S.Orsola Malpighi
Locations (1):
- Azienda Ospedaliero Universitaria Policlinico Sant'Orsola Malpighi, Bologna, BO, Italy